CLINICAL TRIAL: NCT05909228
Title: Bone Turnover Markers in Children With Intestinal Failure After Optimization of Parenteral Nutrition
Brief Title: Bone Markers in Pediatric IF
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000080417
Record Dates: First submitted 2023-05-31; First posted 2023-06-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Intestinal Failure; Osteoporosis; Metabolic Bone Disease
MeSH Terms: conditions — Intestinal Failure; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Bone markers: osteocalcin, bone-specific alkaline phosphatase and c-telopeptide
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with intestinal failure: Children with intestinal failure on parenteral nutrition
- Healthy controls: Healthy controls without parenteral nutrition

SUMMARY:
Poor bone health is a well-recognized but poorly understood complication in children with intestinal failure (IF) who are dependent on parenteral nutrition (PN). Previously, we showed that children with IF have decreased bone turnover markers. It is currently unknown if optimization of parenteral nutrition is related to improved bone turnover markers. Serum concentrations of bone markers (osteocalcin, bone-specific alkaline phosphatase and c-telopeptide) will be measured in 30 IF patients treated at a multidisciplinary intestinal rehabilitation and home PN program at the Hospital for Sick Children and compared to bone markers in 30 age- and sex-matched healthy controls.

DETAILED DESCRIPTION:
It is currently unknown if optimization of PN mixtures leads to a measurable change in bone turnover markers. Our hypothesis is that bone turnover markers of children with IF whose PN has been optimized will not differ from those of healthy control subjects, with a positive effect on bone mineral density.

Our aims are:

* To measure bone turnover markers in children with IF on long-term PN and compare them with age- and sex-matched healthy children who never received PN
* To evaluate if changes in bone turnover markers are related to changes in bone mineral density measured by Dual energy X-ray absorptiometry (DXA)
* To identify IF- and PN-related factors associated with bone health

To be able to answer these aims, bone markers in children with IF will be compared to bone markers in healthy controls, age- and sex-matched.

ELIGIBILITY:
Inclusion criteria are as follows:

In order to be eligible to participate in this study, a patient must meet all of the following criteria at time of inclusion:

1. Consent provided
2. Age < 18 years
3. Suffering from IF needing PN providing at least 25% of calories for ≥6 weeks
4. Medically stable with no acute changes in condition requiring hospitalization, or other intervention at home (for at least 3 months).

For healthy controls the inclusion criteria are as follows:

1. Consent provided
2. Age < 18 years.

A patient who meets any of the following criteria will be excluded from participation in this study:

1. On PN for < 6 weeks
2. Suffering from an acute clinical event, for example gastroenteritis, colds and flu
3. Suffering from sepsis on antibiotics
4. On medication known to affect bone metabolism, for example steroids
5. Having a history of fracture within the last 12 months.

For healthy controls, the exclusion criteria are as follows:

1. Any condition known to affect bone health (chronic disease, bone disease, history of malignancy, radiotherapy, steroid use, mental or physical disability)
2. A positive history of fractures within the past 2 years
3. Poor growth (weight- and height-for-age below - 2 or above + 2 standard deviation score using the WHO growth charts).

Ages: 6 Weeks to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with intestinal failure on parenteral nutrition and healthy controls without parenteral nutrition.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Bone turnover markers - Osteocalcin | Baseline
  To measure serum osteocalcin levels in children with intestinal failure on long-term parenteral nutrition and compare them with age- and sex-matched healthy children who never received parenteral nutrition.
Bone turnover markers - C-telopeptide | Baseline
  To measure serum C-telopeptide levels in children with intestinal failure on long-term parenteral nutrition and compare them with age- and sex-matched healthy children who never received parenteral nutrition.
Bone turnover markers - Bone-specific alkaline phosphatase | Baseline
  To measure serum bone-specific alkaline phosphatase levels in children with intestinal failure on long-term parenteral nutrition and compare them with age- and sex-matched healthy children who never received parenteral nutrition.

SECONDARY OUTCOMES:
Bone health | DXA scan results will be collected when performed within 6 months of the blood draw for the bone markers.
  Association of serum osteocalcin, C-telopeptide and bone-specific alkaline phosphatase with bone mineral density Z-scores for lumber spine and total body less head obtained from DXA scans performed as standard clinical care.
Intestinal failure and parenteral nutrition related factors | Baseline
  Association of intestinal failure and parenteral nutrition related factors such as duration of parenteral nutrition (y) with serum osteocalcin, C-telopeptide and bone-specific alkaline phosphatase levels.
Intestinal failure and parenteral nutrition related factors | Intestinal failure and parenteral nutrition related factors
  Association of intestinal failure and parenteral nutrition related factors such as parenteral nutrition dependency index (%) with serum osteocalcin, C-telopeptide and bone-specific alkaline phosphatase levels.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No